CLINICAL TRIAL: NCT00004181
Title: Allogeneic Bone Marrow Transplantation for Patients With Chronic Myelogenous Leukemia in the Chronic Phase or Multiple Myeloma
Brief Title: Bone Marrow Transplantation in Treating Patients With Multiple Myeloma, Chronic Phase Chronic Myelogenous Leukemia, or Agnogenic Myeloid Metaplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 92H3T; NU-92H3T; NCI-G99-1639
Record Dates: First submitted 2000-01-21; First posted 2003-01-27 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; chronic phase chronic myelogenous leukemia; chronic idiopathic myelofibrosis; Philadelphia chromosome positive chronic myelogenous leukemia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Multiple Myeloma; Neoplasms, Plasma Cell; Leukemia, Myeloid, Chronic-Phase; Primary Myelofibrosis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Busulfan; Cyclophosphamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Procedure: allogeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Bone marrow transplantation may be able to replace immune cells that were destroyed by the chemotherapy or radiation therapy that was used to kill cancer cells.

PURPOSE: Phase II trial to study the effectiveness of allogeneic bone marrow transplantation in treating patients who have multiple myeloma, chronic phase chronic myelogenous leukemia, or agnogenic myeloid metaplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of allogeneic bone marrow transplantation (BMT) following high-dose cyclophosphamide and total body irradiation in patients with multiple myeloma, agnogenic myeloid metaplasia, or chronic myelogenous leukemia in first or second chronic phase.
* Determine the efficacy of BMT following busulfan and cyclophosphamide in these patients.
* Determine the toxic effects of these preparative regimens in these patients.

OUTLINE: Patients are stratified by remission (first vs second vs third).

Patients who have not undergone prior radiotherapy receive cyclophosphamide IV on days -6 and -5 and then undergo total body irradiation twice a day on days -4 to -1. Allogeneic bone marrow is infused on day 0.

Patients who have undergone prior radiotherapy receive oral busulfan every 6 hours on days -7 to -4 or -6 to -3 and cyclophosphamide IV over 2 hours on days -3 and -2. Allogeneic bone marrow is infused on day 0.

Patients are followed at days 30 and 90, at 6 months, and then annually thereafter.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically proven disease of one of the following types with transfusion-dependent anemia or thrombocytopenia (less than 50,000/mm^3):

  * Multiple myeloma
  * Agnogenic myeloid metaplasia
  * Chronic myelogenous leukemia in first or second chronic phase

    * Philadelphia chromosome with BCR gene rearrangement
* Suitable sibling bone marrow donor available

PATIENT CHARACTERISTICS:

Age:

* 15 to physiologic 55

Performance status:

* ECOG 0 or 1

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGOT less than 2 times normal
* Alkaline phosphatase less than 2 times normal

Renal:

* Creatinine less than 2 mg/dL

Cardiovascular:

* Ejection fraction normal by MUGA
* No acute myocardial infarction within the past 6 months
* No active angina pectoris
* No active congestive heart failure

Pulmonary:

* FEV greater than 50% predicted
* DLCO at least 50%

Other:

* HIV negative
* No active infection
* No concurrent organ damage or medical problems that would preclude therapy

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1999-10; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin S. Tallman, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States